CLINICAL TRIAL: NCT02822417
Title: Clinical and Genetic Factors on the Postoperative Recovery Time of General Anaesthesia
Status: Completed | Type: Observational
Sponsor: Yijing He (Other)
Responsible Party: Sponsor-Investigator, Yijing He, Associate professor, Central South University
Organization: Central South University (Other)
Other Study IDs: 2016 MZ/CSU/PS
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: General Anesthesia
Keywords: Recover time

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA retain 1 year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients after general anesthesia: Laparoscopic surgery, orthopedics surgery or open surgery patients after general anesthesia

SUMMARY:
To evaluate the effect of clinical factors on the recovery time of postoperative anesthesia and the effect of genetic variation in gDNA on the recovery time of postoperative anesthesia.

DETAILED DESCRIPTION:
Recovery time of postoperative anesthesia is an important index to reflect patient's postoperative health status. The investigators want to collect patients' clinical dates and their blood samples, then extract DNA from blood samples, acquire every patients' genetic variation information. Finally, acquiring the mathematical model of the influence of clinical factors and genetic factors on the recovery time after operation, predicting the recovery time of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged more than 18 years;
2. General anesthesia for all patients;
3. Patients underwent surgery for laparoscopic surgery, orthopedics surgery or open surgery;
4. Patients were not delivered allogeneic blood in three months;
5. Having the ability to understand and sign the informed consent.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Having an immune deficiency, as a patient with HIV infection;
3. Patients with infectious diseases, such as syphilis;
4. Patients delivered allogeneic blood in three months;
5. Researchers believe that may increasing the risk of subjects or interfering clinical trial;
6. Don't have the ability to understand or sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Laparoscopic surgery, orthopedics surgery or open surgery patients in Chinese
Sampling Method: Probability Sample
Enrollment: 1453 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Recover time of anesthesia | within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yijing He, MD,PhD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
data not entered